CLINICAL TRIAL: NCT01692548
Title: Effect of Neurofeedback Intervention on the Development of ADHD in Children at Risk: a Comparative Study.
Brief Title: Neurofeedback Intervention on the Development of ADHD in Children at Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, larohde, Professor of Chlid and Adolescent Psychiatry, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110084
Record Dates: First submitted 2012-09-12; First posted 2012-09-25 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neurofeedback (Experimental): Neurofeedback: two sessions per week, 30 sessions total.
  Interventions: Other: Neurofeedback
- Control (No Intervention)

INTERVENTIONS:
Other: Neurofeedback
  Arms: Neurofeedback

SUMMARY:
Forty children considered at risk for ADHD (subclinical ADHD) will be randomized to either a neurofeedback intervention or waiting list.

DETAILED DESCRIPTION:
Attention Deficit Hyperactive Disorder (ADHD) is one of the most common mental disorders among children. It is associated with an important burden to individuals, their families and society. ADHD is a chronic condition and the majority of affected individuals presents symptoms and associated functional deficit through adult life. Although pharmacological treatment can be easily implemented and are short-term effective, its efficacy tends to decrease with time and long-term effects are uncertain. Psychosocial treatments tend to be effective only during treatment delivery and treatment effects are not sustained. New treatment strategies are required in order to provide better care to ADHD patients. Early interventions might avoid the development of the disorder, limit its persistency or prevent associated deficits. The aim of this study is to evaluate the efficacy of a non-pharmacological intervention for children at risk for ADHD.

This randomized controlled clinical trial has the aim of testing the efficacy of neurofeedback for children at increased risk for ADHD (subclinical ADHD symptoms). This is study is a multisite school based trial. Forty children from the 1st to the 4th grade with subclinical ADHD symptoms will be randomized to neurofeedback or waiting list. Subclinical ADHD will be defined as having 3-5 out of 9 inattention and/or hyperactivity/impulsivity symptoms according to parents clinical evaluation (K-SADS-PL) but less than 6 symptoms according to teachers report (assessed using SNAP-IV) OR 3-5 symptoms according to teachers report and less than 6 according to parents clinical evaluation. Exclusion criteria includes IQ lower than 80, severe mental disorder or neurological disease. Treatment will comprise 25 sessions of NF using Slow Cortical Potential training. Children will be invited to attend 2 sessions per week, each session comprises 4 blocs of 20 trials with both activation and deactivation challenges. Eldith Tharaprax equipment will be used in both sites. The study, including treatment sessions, will be conducted in schools. Two public schools were selected to host the study, one in São Paulo and another in Porto Alegre, Brazil. Main outcome will be parents rating scores for ADHD symptoms (SWAN questionnaire). To avoid bias due to the low literacy of our population, parents will be assisted by a staff member to fill the SWANs questionnaires. Second outcomes includes: 1) Performance on computerized tests designed to measures time processing, basic processing, inhibitory control and executive function and delay aversion and 2) Pre- post treatment differences on electrophysiological measures (evoke related potentials during two tasks that requires sustained attention, self-monitoring and response to attentional prime); 3) conversion to ADHD (incident cases). Outcomes measures will be assessed prior to treatment start, in after the 13 session, soon after the 25 session, after 6 months of follow-up. Random regression will be used to model each subject's response against time (from baseline to session 12 and from 12th session to treatment end). For continuous variables we will compare the average slope of the regression line across the two groups to test whether the intervention is superior to waiting-list. Proportion of new cases will be compared across groups using chi square test.

ELIGIBILITY:
Inclusion Criteria:

* From 3 to 5 ADHD symptoms according to DSM-IV
* Age 6 to 10

Exclusion Criteria:

* Already attending treatment for ADHD
* IQ below 80

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in ADHD symptoms | Baseline; 6 weeks; 3 months; 6 months.
  Measured by the SWAN scale filled by parents.

SECONDARY OUTCOMES:
Change in performance on computerized tests. | Baseline; 6 weeks; 3 months; 6 months.
  Time processing, basic processing, inhibitory control and executive function and delay aversion.
Change in EEG measures | Baseline; 6 weeks; 3 months; 6 months.
  Pre-post treatment differences on electrophysiological measures (evoke related potentials during two tasks that requires sustained attention, self-monitoring and response to attentional prime)
Incident cases. | 6 months.
  Number of at risk children that actually converts to ADHD diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil